CLINICAL TRIAL: NCT01694082
Title: Randomized, Controlled Trial of a Brief, Web-Based Alcohol Reduction Intervention for Undergraduates
Brief Title: Brief Web-Based Alcohol Reduction Intervention for Undergraduates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Alcoholic Beverage Medical Research Foundation (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Robert Leeman, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1207010596; K01AA019694 (NIH)
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Alcohol Use; Heavy Drinking; Negative Consequences of Alcohol Use
Keywords: brief intervention; web-based interventions; computer-based interventions; harm reduction; young adult; college student
MeSH Terms: conditions — Alcohol Drinking; Harm Reduction | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- THRIVE replication (Experimental): Participants in this condition receive THRIVE with a full list of direct and indirect protective behavioral strategies to reduce alcohol consumption.
  Interventions: Behavioral: THRIVE
- THRIVE direct strategies (Experimental): Participants in this condition receive THRIVE including a subset of protective behavioral strategies that are directly related to alcohol drinking.
  Interventions: Behavioral: THRIVE
- THRIVE indirect strategies (Experimental): Participants in this condition receive THRIVE including a subset of protective behavioral strategies that are indirectly related to alcohol drinking.
  Interventions: Behavioral: THRIVE
- Brief brochure and assessment control (Sham Comparator): Participants will answer the same survey questions as participants in the THRIVE conditions, but will receive a brief alcohol-related brochure with only didactic content rather than the intervention components received by participants randomized to THRIVE conditions.
  Interventions: Behavioral: Brief brochure and assessment control

INTERVENTIONS:
Behavioral: THRIVE — THRIVE stands for (Tertiary Health Research Intervention Via Email). Participants complete questions related to demographics and their alcohol use and receive brief personalized feedback based on this information, in addition to protective behavioral strategies, facts about alcohol and information about available resources to reduce their alcohol use.
  Other Names: Tertiary Health Research Intervention Via Email
  Arms: THRIVE direct strategies; THRIVE indirect strategies; THRIVE replication
Behavioral: Brief brochure and assessment control
  Arms: Brief brochure and assessment control

SUMMARY:
Tertiary Health Research Intervention Via Email (THRIVE; Kypri et al., 2009), originally utilized with Australian students, is unique in that it contains efficacious components derived from motivational interviewing (e.g., personalized feedback) and cognitive behavioral therapy (protective behavioral strategies), yet is very brief and has established efficacy. This study aims to test versions of THRIVE tailored to American college students. In addition to replicating original results with THRIVE, we will also test versions containing unique subsets of protective behavioral strategies to reduce alcohol consumption. The primary hypothesis is that versions of THRIVE will be associated with lower overall alcohol consumption than an assessment and brief brochure control condition.

ELIGIBILITY:
Inclusion Criteria:

* Must be a current student at Albertus Magnus College in New Haven, CT

Exclusion Criteria:

* Under 18 years of age
* 25 years of age or older

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Frequency of alcohol use | 1-month post-intervention
Protective behavioral strategy use | 1-month post-intervention
Overall Weekly Alcohol Consumption | 1-month post-intervention

SECONDARY OUTCOMES:
Frequency of heavy drinking days | 1-month post-intervention
Frequency of alcohol use | 6-months post-intervention
Overall weekly alcohol consumption | 6-months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Leeman, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Frohe T, Gebru NM, Wilson B, Leeman RF. Is a very brief web-based intervention with focus on protective behavioral strategies efficacious in reducing impaired control over alcohol in undergraduates? Exp Clin Psychopharmacol. 2025 Feb;33(1):1-7. doi: 10.1037/pha0000737. Epub 2024 Aug 15. PMID 39146062